CLINICAL TRIAL: NCT04813289
Title: A Retrospective Review of Anaesthetic Practice and Intraoperative Blood Loss in Orthognathic Surgery in a Tertiary Hospital
Brief Title: Review of Anaesthetic Practice in Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/3153
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Maxillofacial Abnormalities; Blood Pressure; Anesthesia
MeSH Terms: conditions — Maxillofacial Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anaesthesia type: 1. Inhalational anaesthesia without Remifentanil use
  2. Inhalational anaesthesia with Remifentanil use
  3. Total intravenous anaesthesia
- Blood pressure monitoring: 1. Intraarterial line use
  2. Non-invasive blood pressure monitoring

SUMMARY:
Orthognathic surgeries for maxillofacial deformities are commonly performed globally. However, they are associated with significant blood loss which can affect the surgical field and result in blood transfusion and its risks. We aim to review the different hypotensive anaesthetic practices for orthognathic surgeries, and their effects on intraoperative blood loss and transfusion requirements.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were scheduled for orthognathic surgeries from January 2014 to March 2017

Exclusion Criteria:

* surgery was not done
* there were missing anaesthetic records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who were scheduled for orthognathic surgeries from January 2014 to March 2017 were included.Patients were excluded from the study if surgery was not done or there were missing anaesthetic records.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Anaesthesia technique | Perioperative
  Most common modality for anaesthesia maintenance

SECONDARY OUTCOMES:
Blood pressure monitoring | Perioperative
  If the use of IA line vs NIBP affected patient outcomes in terms of blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No